CLINICAL TRIAL: NCT03146247
Title: Analysis of the Pathogenesis of Itch in Response to Apremilast Therapy in Psoriasis Patients
Acronym: Itch
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment was not started
Sponsor: Diamant Thaci (Other)
Responsible Party: Sponsor-Investigator, Diamant Thaci, Prof. Dr. med, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C16.Pso-002; 2016-002432-32 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Moderate to Severe Plaque Psoriasis
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (Other): all patients receive same dose and dosing regimen with Apremilast
  Interventions: Drug: Apremilast;Apremilast;Apremilast 10 MG; 20 MG; 30 MG Oral Tablet

INTERVENTIONS:
Drug: Apremilast;Apremilast;Apremilast 10 MG; 20 MG; 30 MG Oral Tablet — All patients are scheduled to receive Apremilast with a titration phase of one week, followed by 23 weeks of regular treatment.

SUMMARY:
This study aims to identify and describe the presence of itch active molecules in psoriasis and response to treatment with apremilast. This data will be complemented by immunohistochemical data determining nerve ending density and neuropeptide concentrations before and during treatment and correlated with patient reported outcome. It is important to underscore that itch may interfere with various aspects of patient functioning, emotions and social status and should therefore be adequately addressed while treating patients with psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand and communicate with the investigator and comply with the requirements of the study and must give written, signed and dated informed consent before any study related activity is performed.
2. Subjects must be at least 18 years of age at time of enrollment
3. Patients with chronic moderate to severe plaque type psoriasis who failed to respond to or who have a contraindication to, or are intolerant to other systemic therapy including cyclosporine, methotrexate or psoralen and ultraviolet-A light (PUVA)
4. Subjects must have a score in the numerical rating scale (NRS, see 12.4) >5 at baseline
5. Women of childbearing potential* and males with female partners of child bearing potential must be ready and able to use highly effective methods of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly.

   * Women of childbearing potential are defined as:

     * Having experienced menarche and
     * not Postmenopausal (12 months with no menses without an alternative medical cause) and
     * not permanently sterilized (e.g. tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)

Exclusion Criteria:

1. Patients with previous treatment with Apremilast
2. Patients incapable of giving full informed consent.Patients enrolled in other clinical trials
3. Allergies against Apremilast or any of the inactive ingredients: lactose monohydrate, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc, iron oxide red, iron oxide yellow (20 and 30 mg only) and iron oxide black (30 mg only)
4. Rifampicin, Phenobarbital, Carbamazepine, Phenytoin, enzalutamid, mitotan or St John's Wort as concomitant medication
5. Patients with rare hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose malabsorption
6. Allergy to local anaesthetic or latex
7. Pregnancy/Lactation
8. Patients with known HIV infection and active or uncontrolled hepatitis B or C infection
9. Patients with known disposition for excessive keloid formation or wound healing disorders
10. Patients with other forms than chronic plaque type psoriasis especially drug-induced psoriasis
11. Patients who cannot tolerate the complete dose used in this study due to medical conditions e.g. due to kidney insufficiency
12. Patients with depressive symptom in PHQ-D in visit 1
13. Concomitant medication that can cause psychiatric symptoms
14. Psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Immunoreactive nerve fibers | until week 16
  Proportion of patients reaching 50% reduction of PGP 9-5- immunoreactive nerve fibers at visit 6 (week 16) compared to visit 1 (week 0) measured with immunohistochemical methods

SECONDARY OUTCOMES:
PASI improvement | until week 16
  Proportion of patients achieving at least 50 % of improvement of PASI at visit 6 (week 16) compared to visit 1 (week 0)

CONTACTS AND LOCATIONS:
Overall Officials: Diamant Thaci, Prof., Principal Investigator — Universität zu Lübeck
Locations (1):
- Comprehensive Center for Inflammation Medicine, UKSH, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No